CLINICAL TRIAL: NCT00687609
Title: An Open Label Pilot Study of Atomoxetine Hydrochloride in Adolescents With Attention Deficit/Hyperactivity Disorder and Comorbid Cannabis Abuse.
Brief Title: Pilot Evaluation of Atomoxetine on Attention Deficit Hyperactivity Disorder (ADHD) Symptoms in Adolescents With Cannabis abusE
Acronym: PEACE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was discontinued early, owing to difficulties in recruiting the target sample after seven patients had been recruited.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12382; B4Z-UT-LYEL (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2010-08-19 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Attention Deficit Hyperactivity Disorder; Cannabis Abuse
Keywords: Attention Deficit Hyperactivity Disorder with Cannabis Abuse; Marihuana Abuse; Comorbid Cannabis Abuse
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Marijuana Abuse | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine (Experimental): 0.5 milligrams per kilogram (mg/kg) daily for 1 week followed by 1.2 mg/kg daily for 11 weeks, orally, capsules.
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — 0.5 milligrams per kilogram (mg/kg) daily for 1 week followed by 1.2 mg/kg daily for 11 weeks, orally, capsules.
  Other Names: LY139603; Strattera

SUMMARY:
The purpose of this study is to determine whether atomoxetine is effective in reducing ADHD (Attention Deficit/Hyperactivity Disorder) symptoms in adolescents with ADHD and comorbid cannabis abuse.

DETAILED DESCRIPTION:
In the past adolescents with cannabis abuse have been excluded from studies in which atomoxetine for ADHD symptoms was studied. In this study the efficacy of atomoxetine on symptoms of ADHD in adolescents with ADHD and comorbid cannabis abuse will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis ADHD based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR)
* At least 1.5 standard deviations above the age norm for their diagnostic subtype using published norms for the ADHD Rating Scale-IV-Parent Version
* Cannabis Abuse or dependence based on the DSM-IV-TR, and using a minimum of 5 joints per week

Exclusion Criteria:

* Weight under 20 kilograms (kg)
* Patients at serious suicidal risk
* Patients with alcohol or drug abuse (other than cannabis)
* Patients who in the investigator's judgement are likely to need psychotropic medication + psychotherapy apart from atomoxetine

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Hague, Netherlands

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was discontinued early owing to difficulties in recruiting the target sample after seven patients had been recruited. Therefore, only disposition, demographic, and safety data are reported.
Period: Overall Study
Arm/Group | Atomoxetine
Started | 7
Completed | 4
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 7
Age Continuous [Mean (Standard Deviation); unit: Years] | 16.3 (0.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 5
  East Asian | 1
  West Asian | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 7
Columbia Suicide Rating Scale (C-SSRS) Suicidal Behavior [Number; unit: Participants] — Solicits suicide-related information with structured questioning. Scale consists of 28 items in 4 sections: suicidal behavior, actual attempts, suicidal ideation, intensity of ideation. Suicidal behavior consists of 7 yes/no items: actual attempt, non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts or behavior, presence of suicidal behavior, completed suicide. Only items with yes responses are listed.
  Participants
    Aborted Attempt | 1
    Non-Suicidal Self Injurious Behavior | 2
    Presence of Suicidal Behavior | 1
    Actual Attempt | 1

OUTCOME MEASURES:

1. Primary Outcome: Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale-IV-Parent Version: Investigator Scored Total Score at 12 Weeks
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54. Higher scores indicate greater impairment. The scale is scored by an investigator while interviewing the parent.
Time Frame: 12 weeks
Population: It was planned to use the full analysis set (FAS) for the efficacy and safety analyses, which included data from all participants who received at least one dose of atomoxetine and had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

2. Secondary Outcome: Clinical Global Impression-ADHD-Improvement (CGI-ADHD-I) at 12 Weeks
Description: Measures total improvement (or worsening) of a patient's ADHD symptoms from the beginning of treatment. (1=very much improved, 7=very much worsened)
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline to 12 Weeks in Global Impression of Perceived Difficulties (GIPD) - Participant Rated Version
Description: The Global Impression of Perceived Difficulties (GIPD) scale is a five-item rating of ADHD-related difficulties. For each item, difficulties during the past week are rated on a 7 point scale (1=normal, not difficult at all; 7= extremely difficult). The GIPD total score is the sum of all subscores (items) and ranges from 5 to 35. Higher scores indicate greater impairment. The scale is completed by the participant.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline to 12 Weeks in the Children's Depression Rating Scale-Revised (CDRS-R)
Description: Measures presence and severity of depression. Consists of 17 items scored on a 1-5 or 1-7 scale (1 = no symptom difficulties; 5 or 7 = severe clinically significant difficulties) A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. In general, scores below 20 indicate an absence of depression; scores of 20 or 30 indicate borderline depression; scores of 40 to 60 indicate moderate depression.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline to 12 Weeks in the Pediatric Anxiety Rating Scale (PARS)
Description: The Pediatric Anxiety Rating Scale (PARS) is used to rate the severity of anxiety in children and adolescents, ages 6 to 17 years. The total score for the PARS is derived by summing 5 of the 7 severity/impairment/interference items (2,3,5,6,7). The total score ranges from 0 (none) to 25 (extreme severity). Items 1 (overall number of anxiety symptoms) and 4 (overall severity of physical symptoms) are not included in the total score calculation.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline to 12 Weeks in the Marijuana Craving Questionnaire (MCQ)
Description: The MCQ is a 12-item self-rated questionnaire to assess cannabis craving with 4 factors: compulsivity (an inability to control marijuana use), emotionality (use of marijuana in anticipation of relief from withdrawal/negative mood), expectancy (anticipation of positive outcomes from smoking marijuana) and purposefulness (intention and planning to use marijuana for positive outcomes). Scores are calculated on a 7-point scale (1=strongly disagree; 7=strongly agree). A separate score is calculated for each factor; scores range from 3-21 each with higher scores indicating greater craving.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Neurocognitive Functioning as Measured at 12 Weeks by a Test Battery: Stop-Signal Task
Description: Consists of 2 types of trials: go trials and stop trials. Go trials require participants to locate the position of an aircraft displayed to the left or right of a fixation point on a computer screen by pressing a left or right button. In 25% of the go stimili an additional stop stimulus (auditory signal) is presented shortly after the go stimulus. Participant then needs to inhibit their response. By varying the time period between go and stop stimulus, 50% of the trials are inhibited successfully, 50% not. The latency of inhibition is estimated. This task takes about 25 minutes.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Neurocognitive Functioning as Measured at 12 Weeks by a Test Battery: Contingency Task
Description: For the Contingency Task participants estimate the duration of a time interval of 1 second by pushing a button. Responses that are within a dynamic time interval are being classified as correct. This way, 50 % of the responses are correct, 50% incorrect. Three contingency conditions: neutral, reward and response cost. The performance of this task takes about 15 minutes.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in Neurocognitive Functioning as Measured at 12 Weeks by a Test Battery: Time Reproduction Task
Description: For the Time Reproduction Task participants need to reproduce the duration of a visual stimulus (lightbulb) by pressing a button. The intervals vary between 2 - 20 seconds. The performance of this task takes about 15 minutes.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Atomoxetine
Number analyzed (Participants) | 0

10. Secondary Outcome: C-SSRS Suicidal Ideation By Visit at Week 4: Non-Specific Active Suicidal Thoughts
Description: Solicits suicide-related information with structured questioning. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, intensity of ideation. Suicidal ideation consists of 5 yes/no items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Only items with yes responses at a given week are listed.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 7
Participants | 1

11. Secondary Outcome: C-SSRS Intensity of Ideation (Most Common Ideation Type and Most Severe Ideation Type) By Visit at Week 4
Description: Participants rate most common and most severe ideation type by frequency (1=<once per week/5=many times/day), duration (1=fleeting/5=>8 times per hour persistent, continuous), controllability (1=easily able to control thoughts/8=no attempt), deterrents to active attempts (1=deterrent definitely stopped you/8=N/A, wish to die only), and reason for ideation (1=completely for attention/revenge/reaction/5=completely to stop the pain). Only items with yes responses at a given week are listed. A participant could have a yes response in more than one item.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 7
Participants
  Frequency (Most Common) Once a Week | 1
  Frequency (Most Severe) Once a Week | 1
  Duration (Most Common) Fleeting | 1
  Duration (Most Severe) Fleeting | 1
  Control (Most Common) Little Diffficulty | 1
  Control (Most Severe) Little Diffficulty | 1
  Deterrent (Most Common) Uncertain It Stopped You | 1
  Deterrent (Most Severe) Uncertain it Stopped You | 1
  Reasons (Most Common) Mostly to Get Attention | 1
  Reasons (Most Severe) Mostly to Get Attention | 1

ADVERSE EVENTS:
Arm/Group | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=7)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Irritability (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Decreased activity (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The study was discontinued early, owing to difficulties in recruiting the target sample after seven patients had been recruited. Therefore, only disposition, demographic, and safety data are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days